CLINICAL TRIAL: NCT02228564
Title: A Prospective, Multi-Center, Non-Randomized, Single-Arm Study of the BARD® LIFESTREAM™ Balloon Expandable Vascular Covered Stent in the Treatment of Iliac Artery Occlusive Disease (BOLSTER)
Brief Title: BARD® Study of LIFESTREAM™ Balloon Expandable Covered Stent Treating Iliac Arterial Occlusive Disease
Acronym: BOLSTER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: C. R. Bard (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BPV-12-001
Record Dates: First submitted 2014-08-15; First posted 2014-08-29 (Estimated); Results first posted 2020-10-08 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-09

CONDITIONS: Peripheral Artery Disease; Peripheral Vascular Disease; Arterial Occlusive Disease
Keywords: Lack of perfusion in the extremities; Atherosclerosis; Intermittent claudication; BOLSTER
MeSH Terms: conditions — Peripheral Arterial Disease; Peripheral Vascular Diseases; Arterial Occlusive Diseases; Atherosclerosis; Intermittent Claudication | interventions — Angioplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: Yes

ARMS (1):
- LIFESTREAM™ (Experimental): This is a single arm study. All subjects receive percutaneous transluminal angioplasty (PTA) and implantation of the LIFESTREAM™ covered stent.
  Interventions: Procedure: Percutaneous transluminal angioplasty (PTA); Device: LIFESTREAM™ covered stent

INTERVENTIONS:
Procedure: Percutaneous transluminal angioplasty (PTA) — Percutaneous transluminal angioplasty (PTA) is a procedure that can open up a blocked blood vessel using a small, flexible plastic tube, or catheter, with a "balloon" at the end of it. When the tube is in place, it inflates to open the blood vessel, or artery, so that normal blood flow is restored.
Device: LIFESTREAM™ covered stent — Implantation of the LIFESTREAM™ covered stent

SUMMARY:
Collect confirmatory evidence of the safety and effectiveness of the Balloon LIFESTREAM™ Stent Graft for the treatment of stenoses and occlusion in the iliac arteries.

ELIGIBILITY:
CLINICAL INCLUSION CRITERIA:

* The subject provides written informed consent using an Informed Consent Form approved by the Ethics Committee/ Institutional Review Board for the site.
* Subject agrees to comply with the protocol-mandated follow-up procedures and visits.
* Subject is a male or non-pregnant female ≥ 21 years old with an expected lifespan sufficient to allow for completion of all study procedures.
* Subject has intermittent claudication (Rutherford Category 2-3) or ischemic rest pain (Rutherford Category 4).
* Subject is able and willing to comply with any required medication regimen.

ANGIOGRAPHIC INCLUSION CRITERIA:

* Subject has evidence of single, bilateral, or multiple de novo and/or restenotic (non-stented) lesion in the native common and/or external iliac artery that is ≥ 50% stenosed (including total occlusions).
* The target lesion can be successfully crossed with a guide wire and pre-dilated with an appropriately sized PTA balloon.
* The reference vessel diameter is between 4.5 mm -12.0 mm in diameter.
* The target lesion is ≤ 100 mm in combined length (per side).
* The subject has angiographic evidence of a patent (< 50% stenosis) profunda and/or superficial femoral artery (SFA) in the target limb.

CLINICAL EXCLUSION CRITERIA:

* The subject is unable or unwilling to provide written informed consent or to conform to the study protocol follow-up procedures and visits.
* The subject is or plans to become pregnant during the study.
* The subject is asymptomatic, has mild claudication or critical limb ischemia with tissue loss described as Rutherford Category 0, 1, 5 or 6.
* The subject has a vascular graft previously implanted in the native iliac vessel.
* The subject suffered a hemorrhagic stroke or transient ischemic attack (TIA) within 3 months prior to the index procedure.
* The subject has a known uncorrectable bleeding diathesis or active coagulopathy.
* The subject has a serum creatinine ≥ 2.5 mg/dl or is on dialysis.
* The subject has a known allergy or sensitivity to stainless steel (i.e., Nickel), ePTFE, or has intolerance to the antiplatelet, anticoagulant or thrombolytic medications required per the protocol.
* The subject has a known allergy or sensitivity to contrast media, which cannot be adequately pre-medicated.
* The subject had a prior vascular intervention within 30 days before or planned for within 30 days after the index procedure.
* The subject has another medical condition, which may cause him/her to be non-compliant with the protocol, confound the data interpretation, or is associated with a life expectancy insufficient to allow for the completion of study procedures and follow-up.
* The subject is currently participating in an investigational drug, biologic, or another device study.

ANGIOGRAPHIC EXCLUSION CRITERIA:

* The subject has extensive peripheral vascular disease, which in the opinion of the Investigator, would preclude safe insertion of an introducer sheath. The ipsilateral common femoral artery should be patent (< 50% stenosis).
* The target lesion requires treatment other than angioplasty to facilitate subject device delivery.
* The subject has severe calcification of the target lesion, preventing inflation of PTA balloon.
* The target lesion has been previously treated with a stent (bare or covered).
* The subject has angiographic evidence of acute thrombus at the target lesion.
* The target lesion involves the origin of the internal iliac artery such that successful treatment of the lesion would require the subject device to cross/occlude the side branch.
* The target lesion located in the distal external iliac artery such that successful treatment of the lesion would require the subject device to cross/occlude side branches or be exposed to compressive forces associated with the close proximity to the common femoral artery.
* The subject has an abdominal aortic aneurysm (AAA) contiguous to the iliac artery target lesion.
* The subject has a pre-existing target iliac artery aneurysm or perforation or dissection of the target iliac artery prior to the initiation of the treatment for this study.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2014-09; Primary Completion 2016-12 (Actual); Study Completion 2018-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John R Laird, M.D., Principal Investigator — U. C. Davis Medical Center
Locations (20):
- United States (14):
  - Arkansas Heart Hospital, Little Rock, Arkansas
  - Vascular and Interventional Specialists of Orange County, Orange, California
  - UC Davis Cardiovascular Medicine, Sacramento, California
  - Florida Research Network, Gainesville, Florida
  - Baptist Medical Center, Jacksonville, Florida
  - Lakeland Regional Medical Center, Lakeland, Florida
  - Mount Sinai Medical Center, Miami, Florida
  - University of Massachusetts Worcester, Worcester, Massachusetts
  - Kansas City Vascular Foundation, Kansas City, Missouri
  - CaroMont Regional Medical Center, Gastonia, North Carolina
  - North Carolina Heart and Vascular, Raleigh, North Carolina
  - Donald Guthrie Foundation, Sayre, Pennsylvania
  - Univeristy of Texas Medical Branch, Galveston, Texas
  - Swedish Health Services, Seattle, Washington
- Germany (5):
  - Universitäts-Herzzentrum Freiburg-Bad Krozingen GmbH, Bad Krozingen
  - Ev.Krankenhaus Königin Elisabeth, Berlin
  - Praxis fur Interventionelle Angiologie, Kaiserslautern
  - Universitaetsklinikum Leipzig, Leipzig
  - Bonifatius Hospital, Lingen
- Auckland Hospital, Auckland, New Zealand

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | LIFESTREAM™
Started | 155
Completed | 106
Not Completed | 49
Not completed — Withdrawal by Subject | 10
Not completed — Death | 11
Not completed — Physician Decision | 5
Not completed — Lost to Follow-up | 17
Not completed — Other | 6

BASELINE CHARACTERISTICS:
Arm/Group | LIFESTREAM™
Number analyzed (Participants) | 155
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.3 (9.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48
  Male | 107
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 150
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  New Zealand | 21
  United States | 57
  Germany | 77

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Device and/or Procedure-Related Death or Myocardial Infarction (MI) Through 30 Days, or Any Target Lesion Revascularization (TLR), Target Limb(s) Major Amputation, or Restenosis Through 9-Months Post Index Procedure.
Description: The primary endpoint is a composite safety and effectiveness measure defined as device and/or procedure-related death or myocardial infarction (MI) through 30 days, or any Target Lesion Revascularization (TLR), target limb(s) major amputation, or restenosis through 9-months post-index procedure.
Time Frame: 9 months post index procedure
Population: The number of participants (n) may vary from the total number of participants (N) in the study as n depends on the number of participants for which data was available at the given time-point analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | LIFESTREAM™
Number analyzed (Participants) | 138
Participants | 16
Statistical Analysis 1: Comparison: LIFESTREAM™; H0: The proportion of subjects in the LifeStream™ Covered Stent group (PBBX) with events in the primary endpoint is greater than or equal to that of the PG of 19.5%. H1: The proportion of subjects in the LifeStream™ Covered Stent group (PBBX) with events in the primary endpoint is less than that of the PG of 19.5%; Test type: Non-Inferiority — The sample size calculation assumes the following: The LIFESTREAM™ Covered Stent composite event rate is estimated at 10.5% The Performance Goal is set at 19.5% The Type 1 error, α = 0.05 (one-sided). The Type 2 error, β = 0.10 (Power = 1 - β = 90%). The calculated sample size is 139 subjects to be followed through the 9-month follow-up visit (using nQuery 7.0). To accommodate 10% censoring, the sample size is increased to 154; p < 0.0325, Exact binomial test

2. Secondary Outcome: Number of Participants With Major Adverse Events (MAEs) Through 9-Months Post Index Procedure.
Description: Major Adverse Events (MAE) defined as device and/or procedure-related death or MI through 30 days, or any TLR or target limb(s) major amputation through 9-months post-index procedure. Major amputation is defined as an amputation at or above the ankle.
Time Frame: 9 months post index procedure
Population: The number of participants (n) varies from the total number of participants (N) in the study as n depends on the number of participants for which data was available at the given time-point analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | LIFESTREAM™
Number analyzed (Participants) | 150
Participants | 7

3. Secondary Outcome: Number of Lesions With Acute Lesion Success
Description: Acute Lesion Success defined as attainment of < 30% residual stenosis of the target lesion after the index procedure using any percutaneous method and/or non-investigational device (i.e., post-dilatation), as determined by an Independent Angiographic Core Lab.
Time Frame: At time of Index Procedure
Measure: Count of Units; unit: Lesions
Units Other Than Participants: Lesions
Arm/Group | LIFESTREAM™
Number analyzed (Participants) | 155
Number analyzed (Lesions) | 191
Lesions | 188

4. Secondary Outcome: Number of Participants With Acute Procedure Success
Description: Acute Procedure Success defined as lesion success and no peri-procedural complications (death, stroke, myocardial infarction (MI), emergent surgical revascularization, significant distal embolization in target limb, and thrombosis of target vessel) prior to hospital discharge.
Time Frame: At time of hospital discharge
Population: The number of participants (n) varies from the total number of participants (N) in the study as n depends on the number of participants for which data was available at the given time-point analysis. In this instance, three subjects did not have procedure angiography data.
Measure: Count of Participants; unit: Participants
Arm/Group | LIFESTREAM™
Number analyzed (Participants) | 152
Participants | 148

5. Secondary Outcome: Number of Devices With Acute Technical Success at Index Procedure
Description: Acute Technical Success defined as successful deployment of the LIFESTREAM™ Covered Stent at the intended location, as determined by the Investigator.
Time Frame: At time of index procedure
Measure: Count of Units; unit: Devices
Units Other Than Participants: Devices
Arm/Group | LIFESTREAM™
Number analyzed (Participants) | 155
Number analyzed (Devices) | 230
Devices | 226

6. Secondary Outcome: Number of Participants With Target Lesion Revascularization (TLR) at 6, 9, 12, 24, and 36 Months Post Index Procedure
Description: Target Lesion Revascularization (TLR) is defined as the first revascularization procedure (e.g., PTA, atherectomy, etc.) of the target lesion(s) following the index procedure, as determined by an Independent Angiographic Core Lab. All Target Lesion Revascularizations (TLR) were Target Vessel Revascularizations (TVR) and therefore, the results presented in Outcome #6 and Outcome #7 are the same.
Time Frame: 6, 9, 12, 24, and 36 months post index procedure
Population: The number of participants analyzed (n) at each time point varies from the total of participants in the study (N) in relation to subjects censored at each time point.
Measure: Number; unit: Participants
Arm/Group | LIFESTREAM™
Number analyzed (Participants) | 155
Participants
  6 months post index procedure: number analyzed (Participants) | 154
  6 months post index procedure | 3
  9 months post index procedure: number analyzed (Participants) | 149
  9 months post index procedure | 5
  12 months post index procedure: number analyzed (Participants) | 146
  12 months post index procedure | 7
  24 months post index procedure: number analyzed (Participants) | 137
  24 months post index procedure | 19
  36 Months Post Index Procedure: number analyzed (Participants) | 89
  36 Months Post Index Procedure | 23

7. Secondary Outcome: Number of Participants With Target Vessel Revascularization (TVR) Event at 6, 9, 12, 24, and 36 Months Post Index Procedure.
Description: Target Vessel Revascularization (TVR) is defined as the first revascularization procedure (e.g. PTA, stenting, surgical bypass, etc.) in the target vessel(s) following the index procedure, as determined by an Independent Angiographic Core Lab. All Target Vessel Revascularizations (TVR) were Target Lesion Revascularizations (TLR) and therefore, the results presented in Outcome #6 and Outcome #7 are the same.
Time Frame: 6, 9, 12, 24, and 36 months post index procedure
Population: as for outcome 6
Measure: Number; unit: Participants
Arm/Group | LIFESTREAM™
Number analyzed (Participants) | 155
Participants
  6 months post index procedure: number analyzed (Participants) | 154
  6 months post index procedure | 3
  9 months post index procedure: number analyzed (Participants) | 149
  9 months post index procedure | 5
  12 months post index procedure: number analyzed (Participants) | 146
  12 months post index procedure | 7
  24 months post index procedure: number analyzed (Participants) | 137
  24 months post index procedure | 19
  36 Months Post Index Procedure: number analyzed (Participants) | 89
  36 Months Post Index Procedure | 23

8. Secondary Outcome: Number of Participants With Sustained Clinical Success at 30-Days and 9, 12, 24, and 36 Months Post Index Procedure
Description: Sustained Clinical Success defined as sustained cumulative improvement from baseline value of ≥ 1 Rutherford Category23 at 30-days and 9, 12, 24, and 36-months post-index procedure, as determined by the Investigator.
Time Frame: 30 days, and 9, 12, 24, and 36 months post index procedure
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | LIFESTREAM™
Number analyzed (Participants) | 155
Participants
  30 days post index procedure: number analyzed (Participants) | 150
  30 days post index procedure | 133
  9 months post index procedure: number analyzed (Participants) | 137
  9 months post index procedure | 124
  12 months post index procedure: number analyzed (Participants) | 132
  12 months post index procedure | 124
  24 months post index procedure: number analyzed (Participants) | 117
  24 months post index procedure | 106
  36 months post index procedure: number analyzed (Participants) | 106
  36 months post index procedure | 98

9. Secondary Outcome: Number of Participants With Primary Patency at 9, 12, 24, and 36 Months Post Index Procedure
Description: Primary Patency at 9, 12, 24 and 36-months post-index procedure corresponding to PSVR ≤ 2.4.
Time Frame: 9, 12, 24 and 36 months post index procedure
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | LIFESTREAM™
Number analyzed (Participants) | 155
Participants
  9 months post index procedure: number analyzed (Participants) | 138
  9 months post index procedure | 118
  12 months post index procedure: number analyzed (Participants) | 133
  12 months post index procedure | 110
  24 months post index procedure: number analyzed (Participants) | 121
  24 months post index procedure | 92
  36 months post index procedure: number analyzed (Participants) | 105
  36 months post index procedure | 72

10. Secondary Outcome: Number of Participants With Assisted Primary Patency at 9, 12, 24, and 36 Months Post Index Procedure
Description: Primary Assisted Patency at 9-, 12-, 24-, and 36-months post-index procedure corresponding to PSVR ≤ 2.4, as determined by an Independent DUS Core Lab. Primary Assisted Patency is independent of whether or not patency is re-established via an endovascular procedure following restenosis.
Time Frame: 9, 12, 24, and 36 months post index procedure
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | LIFESTREAM™
Number analyzed (Participants) | 155
Participants
  9 months post index procedure: number analyzed (Participants) | 138
  9 months post index procedure | 119
  12 months post index procedure: number analyzed (Participants) | 132
  12 months post index procedure | 112
  24 months post index procedure: number analyzed (Participants) | 117
  24 months post index procedure | 98
  36 months post index procedure: number analyzed (Participants) | 99
  36 months post index procedure | 78

11. Secondary Outcome: Number of Participants With Secondary Patency at 9, 12, 24, and 36 Months Post Index Procedure.
Description: Secondary Patency is a measure of success at re-establishing patency following failure of the initial stent placement due to stenosis or re-occlusion. In this study, Secondary Patency was independent of whether or not patency was re-established via an endovascular procedure following restenosis or occlusion, and was analyzed for the Intent to Treat (ITT) population. Secondary patency is defined as a peak systolic velocity ratio (PSVR) ≤ 2.4, as determined by an independent Duplex Ultrasonography (DUS) Core Lab.
Time Frame: 9,12, 24, and 36 months post index procedure
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | LIFESTREAM™
Number analyzed (Participants) | 137
Participants
  9 months post index procedure | 121
  12 months post index procedure: number analyzed (Participants) | 129
  12 months post index procedure | 112
  24 months post index procedure: number analyzed (Participants) | 113
  24 months post index procedure | 100
  36 months post index procedure: number analyzed (Participants) | 91
  36 months post index procedure | 79

12. Secondary Outcome: Change in Walking Impairment Questionnaire (WIQ) Scores at 30 Days, 9, 12, 24, and 36-Months Post Index Procedure Compared to Baseline.
Description: The WIQ assesses 3 categories of activities that include 1) walking distance, 2) stair-climbing, and 3) walking speed. Each question requires participants to rate their degree of difficulty with the activity on a scale of 0 (unable) to 4 (no problem). Final scores range from 0% to 100%, with lower percentages indicating higher levels of difficulties with activities.The results below represent the mean differences in total Walking Impairment Questionnaire (WIQ) scores at 30 days,9, 12, 24, and 36 months compared to baseline assessment scores.
Time Frame: 30 Days, 9, 12, 24, and 36 months post index procedure compared to baseline.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | LIFESTREAM™
Number analyzed (Participants) | 155
Score on a scale
  30-days Post Index Procedure: number analyzed (Participants) | 148
  30-days Post Index Procedure | 31.45 (25.23)
  9 months post index procedure: number analyzed (Participants) | 134
  9 months post index procedure | 32.10 (26.84)
  12 months post index procedure: number analyzed (Participants) | 130
  12 months post index procedure | 32.81 (26.75)
  24 months post index procedure: number analyzed (Participants) | 116
  24 months post index procedure | 31.34 (26.77)
  36 Months Post Index Procedure: number analyzed (Participants) | 103
  36 Months Post Index Procedure | 32.52 (27.27)

ADVERSE EVENTS:
Arm/Group | LIFESTREAM™
All-Cause Mortality (participants affected / at risk) | 11/155
Serious Adverse Events (participants affected / at risk) | 60/155
Other Adverse Events (participants affected / at risk) | 134/155
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LIFESTREAM™ (N=155)
Anaemia (Blood and lymphatic system disorders) | 3
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Acute Coronary Syndrome (Cardiac disorders) | 1
Acute Myocardial Infarction (Cardiac disorders) | 5
Aortic Valve Stenosis (Cardiac disorders) | 1
Atrial Fibrillation (Cardiac disorders) | 5
Atrioventricular Block Complete (Cardiac disorders) | 1
Bradycardia (Cardiac disorders) | 1
Cardiac Arrest (Cardiac disorders) | 2
Cardiac Failure (Cardiac disorders) | 2
Cardiac Failure Congestive (Cardiac disorders) | 4
Cardiogenic Shock (Cardiac disorders) | 1
Cardiomyopathy (Cardiac disorders) | 1
Coronary Artery Disease (Cardiac disorders) | 3
Coronary Artery Occlusion (Cardiac disorders) | 1
Myocardial Infarction (Cardiac disorders) | 1
Pericardial Effusion (Cardiac disorders) | 1
Ventricular Tachycardia (Cardiac disorders) | 1
Vestibular Disorder (Ear and labyrinth disorders) | 1
Cataract (Eye disorders) | 1
Retinal Vein Thrombosis (Eye disorders) | 1
Abdominal Discomfort (Gastrointestinal disorders) | 1
Duodenal Ulcer (Gastrointestinal disorders) | 1
Gastric Ulcer (Gastrointestinal disorders) | 1
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 3
Inguinal Hernia (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Pancreatitis Chronic (Gastrointestinal disorders) | 1
Retroperitoneal Haemorrhage (Gastrointestinal disorders) | 1
Small Intestinal Obstruction (Gastrointestinal disorders) | 2
Adverse Drug Reaction (General disorders) | 1
Chest Pain (General disorders) | 1
Death (General disorders) | 1
Device Occlusion (General disorders) | 8
Non-Cardiac Chest Pain (General disorders) | 1
Thrombosis In Device (General disorders) | 2
Vessel Puncture Site Bruise (General disorders) | 1
Cholecystitis Chronic (Hepatobiliary disorders) | 1
Gallbladder Perforation (Hepatobiliary disorders) | 1
Bacteraemia (Infections and infestations) | 1
Bronchopneumonia (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Cholecystitis Infective (Infections and infestations) | 1
Diverticulitis (Infections and infestations) | 2
Gangrene (Infections and infestations) | 1
Groin Abscess (Infections and infestations) | 1
Haematoma Infection (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Kidney Infection (Infections and infestations) | 1
Osteomyelitis (Infections and infestations) | 1
Perirectal Abscess (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 1
Scrotal Abscess (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Septic Shock (Infections and infestations) | 1
Subcutaneous Abscess (Infections and infestations) | 1
Urosepsis (Infections and infestations) | 3
Ankle Fracture (Injury, poisoning and procedural complications) | 1
Laceration (Injury, poisoning and procedural complications) | 1
Peripheral Arterial Reocclusion (Injury, poisoning and procedural complications) | 2
Peripheral Artery Restenosis (Injury, poisoning and procedural complications) | 9
Pneumothorax Traumatic (Injury, poisoning and procedural complications) | 1
Postoperative Ileus (Injury, poisoning and procedural complications) | 1
Radial Nerve Injury (Injury, poisoning and procedural complications) | 1
Thermal Burn (Injury, poisoning and procedural complications) | 1
Toxicity To Various Agents (Injury, poisoning and procedural complications) | 1
Vascular Graft Occlusion (Injury, poisoning and procedural complications) | 1
Vascular Pseudoaneurysm (Injury, poisoning and procedural complications) | 3
Wound (Injury, poisoning and procedural complications) | 1
Wrist Fracture (Injury, poisoning and procedural complications) | 1
Haemoglobin Decreased (Investigations) | 1
Staphylococcus Test (Investigations) | 1
Abnormal Loss Of Weight (Metabolism and nutrition disorders) | 1
Diabetes Mellitus Inadequate Control (Metabolism and nutrition disorders) | 1
Failure To Thrive (Metabolism and nutrition disorders) | 1
Fluid Overload (Metabolism and nutrition disorders) | 2
Hyponatraemia (Metabolism and nutrition disorders) | 1
Malnutrition (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Compartment Syndrome (Musculoskeletal and connective tissue disorders) | 1
Immune-Mediated Necrotising Myopathy (Musculoskeletal and connective tissue disorders) | 1
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2
Rotator Cuff Syndrome (Musculoskeletal and connective tissue disorders) | 2
Spinal Column Stenosis (Musculoskeletal and connective tissue disorders) | 1
Spinal Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2
Bladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Brain Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Colon Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hepatocellular Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant Neoplasm Of Pleura (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Squamous Cell Carcinoma Of Lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Carotid Artery Occlusion (Nervous system disorders) | 1
Carotid Artery Stenosis (Nervous system disorders) | 7
Cerebellar Ischaemia (Nervous system disorders) | 1
Cervical Myelopathy (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Presyncope (Nervous system disorders) | 1
Radial Nerve Palsy (Nervous system disorders) | 1
Sciatica (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Transient Ischaemic Attack (Nervous system disorders) | 3
Psychosomatic Disease (Psychiatric disorders) | 1
Bladder Mass (Renal and urinary disorders) | 2
Calculus Urinary (Renal and urinary disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 2
Renal Artery Stenosis (Renal and urinary disorders) | 1
Renal Failure (Renal and urinary disorders) | 1
Renal Failure Acute (Renal and urinary disorders) | 5
Urethral Stenosis (Renal and urinary disorders) | 1
Urinary Retention (Renal and urinary disorders) | 3
Cervical Dysplasia (Reproductive system and breast disorders) | 1
Genital Prolapse (Reproductive system and breast disorders) | 1
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 1
Incisional Drainage (Surgical and medical procedures) | 1
Arteriovenous Fistula (Vascular disorders) | 1
Diabetic Microangiopathy (Vascular disorders) | 1
Hypertensive Crisis (Vascular disorders) | 1
Iliac Artery Occlusion (Vascular disorders) | 1
Intermittent Claudication (Vascular disorders) | 1
Leriche Syndrome (Vascular disorders) | 1
Peripheral Arterial Occlusive Disease (Vascular disorders) | 14
Peripheral Artery Dissection (Vascular disorders) | 1
Peripheral Artery Stenosis (Vascular disorders) | 19
Peripheral Artery Thrombosis (Vascular disorders) | 2
Peripheral Embolism (Vascular disorders) | 1
Peripheral Ischaemia (Vascular disorders) | 2
Subclavian Artery Occlusion (Vascular disorders) | 1
Subclavian Artery Stenosis (Vascular disorders) | 1
Venous Insufficiency (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LIFESTREAM™ (N=155)
Atrial Fibrillation (Cardiac disorders) | 8
Adverse Drug Reaction (General disorders) | 9
Device Occlusion (General disorders) | 8
Oedema Peripheral (General disorders) | 8
Vessel Puncture Site Haematoma (General disorders) | 9
Peripheral Artery Restenosis (Injury, poisoning and procedural complications) | 17
Carotid Artery Stenosis (Nervous system disorders) | 11
Renal Failure Acute (Renal and urinary disorders) | 9
Peripheral Arterial Occlusive Disease (Vascular disorders) | 19
Peripheral Artery Dissection (Vascular disorders) | 9
Peripheral Artery Stenosis (Vascular disorders) | 39

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Prior to PI publication of site results, sponsor requires publication of multi-centers results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-06-15): https://cdn.clinicaltrials.gov/large-docs/64/NCT02228564/Prot_SAP_000.pdf